CLINICAL TRIAL: NCT01309880
Title: A Study to Evaluate the Product Feasibility of a New Silicone Hydrogel Contact Lens
Brief Title: Evaluation of a New Silicone Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 686E
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Myopia
Keywords: Contact lens
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air Optix Aqua (Active Comparator): Ciba Vision daily wear contact lens
  Interventions: Device: Air Optix Aqua
- Test Lens (Experimental): Investigational silicone hydrogel contact lens
  Interventions: Device: Test lens

INTERVENTIONS:
Device: Test lens — Investigational silicone hydrogel contact lens worn on a daily wear basis
  Arms: Test Lens
Device: Air Optix Aqua — Air Optix Aqua contact lens worn on a daily wear basis
  Arms: Air Optix Aqua

SUMMARY:
The objective of this study is to determine the clinical feasibility and to evaluate the product performance of investigational contact lenses developed by Bausch + Lomb.

ELIGIBILITY:
Inclusion Criteria:

* Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
* Be adapted wearers of soft contact lenses, wear a lens in each eye, and each lens must be of the same manufacture and brand.

Exclusion Criteria:

* Have worn gas permeable (GP) contact lenses within last 30 days or polymethylmethacrylate (PMMA) lenses within last 3 months.
* Any systemic disease affecting ocular health.
* Using any systemic or topical medications that will affect ocular physiology or lens performance.
* An active ocular disease, any corneal infiltrative response or are using any ocular medications.
* Any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Allergic to any component in the study care products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-12; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Barna, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a randomized, bilateral, subject-masked, two-week study with a crossover at one week, conducted at three sites in the United States (US). First participant was enrolled on 12/01/2010, last participant exited the study on 12/23/2010.
Pre-assignment Details: A total of 66 participants (132 eyes) were enrolled in the study. One-half (33) were randomized to receive the investigational RD2117-01 ID4 contact lens first, and the other half (33) was randomized to receive the Air Optix Aqua contact lens first then crossed over after 1 week. All participants completed the study.
Groups:
- Air Optix Aqua Then Test Lens: Ciba Vision Air Optix Aqua contact lens. Lenses were worn on a daily wear basis. After one week participants crossed over to the Test lens. All subjects were provided with Bausch + Lomb renu® fresh™ multi-purpose solution and lens cases for daily rinsing, cleaning, disinfecting, and storing their lenses, and Bausch + Lomb Sensitive Eyes® Rewetting Drops for use as needed during the study.
- Test Lens Then Air Optix Aqua: The test lens was an Investigational silicone hydrogel contact lens. Lenses were worn on a daily wear basis. After one week participants crossed over to Ciba Vision Air Optix Aqua contact lens.. All subjects were provided with Bausch + Lomb renu® fresh™ multi-purpose solution and lens cases for daily rinsing, cleaning, disinfecting, and storing their lenses, and Bausch + Lomb Sensitive Eyes® Rewetting Drops for use as needed during the study.
Period: Overall Study
Arm/Group | Air Optix Aqua Then Test Lens | Test Lens Then Air Optix Aqua
Started | 33 | 33
Completed | 33 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All eligible enrolled participants
Groups:
- Overall Study: One-half of the participants (33) were randomized to receive the investigational RD2117-01 ID4 contact lens, and the other half (33) was randomized to receive the Air Optix Aqua contact lens. Both groups wore the lenses on a daily wear basis. After one week of wearing the first lens type, the subjects returned for an exam and crossed over to the second lens type for one week.
Arm/Group | Overall Study
Number analyzed (Participants) | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 66

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Distance high contrast logMAR lens visual acuity (VA) between the Air Optix Aqua lens and the Test Lens at Dispensing and at 1-Week Follow-up.
Time Frame: Dispensing & 1-week follow up
Population: All Eligible, Dispensed Eyes
Measure: Least Squares Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Air Optix Aqua | Test Lens
Number analyzed (Participants) | 66 | 66
Number analyzed (eyes) | 132 | 132
logMAR
  Dispensing | -0.083 (0.071) | -0.085 (0.071)
  1-Week Follow-up | -0.084 (0.077) | -0.078 (0.077)

2. Secondary Outcome: Slit Lamp Findings
Description: Measured on a scale of 0-4 where 0=none, 1=trace, 2=mild, 3=moderate, and 4=severe for edema, microcysts, corneal staining, limbal injection, bulbar injection, upper lid tarsal conjunctival abnormalities, corneal neovascularization and corneal infiltrates.
Time Frame: 1 week
Population: All Dispensed Eyes
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Air Optix Aqua | Test Lens
Number analyzed (Participants) | 66 | 66
Number analyzed (eyes) | 132 | 132
eyes
  Grade 0 | 46 | 82
  Grade 1 | 86 | 50
  Grade 2 | 0 | 0
  > Grade 2 | 0 | 0

3. Secondary Outcome: Comfort
Description: At 1-Week Follow-up, participants rated lens comfort on a scale of 0 to 100, with 100 being the most favorable score.
Time Frame: 1 Weeks
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Air Optix Aqua | Test Lens
Number analyzed (Participants) | 66 | 66
Number analyzed (eyes) | 132 | 132
units on a scale | 85.5 (19.5) | 81.8 (19.5)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Air Optix Aqua | Test Lens
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 0/66 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other